CLINICAL TRIAL: NCT00393107
Title: Phase II Study of Rituximab in Combination With Fludarabine and Cyclophosphamide for the Treatment of Relapsed Follicular Lymphoma
Brief Title: Safety and Efficacy of Fludarabine and Cyclophosphamide + Rituximab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Studio Linfomi (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FR2; FolRec02; GislFR2
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2006-10-26 (Estimated); Status verified 2006-10

CONDITIONS: Follicular Lymphoma
Keywords: follicular lymphoma; non-Hodgkin lymphoma; Fludarabine; Cyclophosphamide; Rituximab; combination; immuno-chemotherapy; relapsed
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Recurrence | interventions — Rituximab; fludarabine; Cyclophosphamide

INTERVENTIONS:
Drug: rituximab
Drug: rituximab,fludarabine, cyclophosphamide

SUMMARY:
Purpose of this study was to assess the safety profile and the anti-lymphoma activity of the FC+R combination.

DETAILED DESCRIPTION:
The natural history of follicular lymphomas is characterized by a high initial response rate to chemotherapy followed invariably by relapse, with subsequent remissions of progressively shorter duration. The majority of patients eventually die of their disease. As yet, there is no gold standard for the treatment of newly diagnosed or relapsed advanced FL.Rituximab(R) has been shown to be a highly effective agent in the treatment of FL, either alone or in combination with chemotherapy. The ability of R to sensitize indolent lymphoma derived cell lines to cytotoxic chemotherapy agents has been demonstrated. Furthermore, fludarabine (F) may also sensitize cells to the effects of R. Cyclophosphamide (C) and F have shown in vivo synergistic activity. In view of the single agent activity and demonstrated synergy between C and F, and between F and R, we evaluated FC+R in previously treated patients with advanced FL. The primary aim of this study was to assess the safety profile and clinical activity of the FC+R combination. The secondary goal was to evaluate the ability of the treatment to convert bone marrow Bcl2 positivity such that patients achieved molecular remissions.

ELIGIBILITY:
Inclusion Criteria:

* histologically documented WHO grade 1-2 ,CD20+,follicular lymphoma
* relapsed Follicular lymphoma
* stage III or IV disease
* Stage II patients are eligible if they present with B symptoms or bulky disease
* to have a need for therapy in the opinion of treating clinician
* measurable disease
* expected survival of 6 months or more
* age 18 to 70 years
* to have undergone < 3 lines of chemotherapy
* performance status of 0 to 2

Exclusion Criteria:

* known HIV infections
* Known Hepatitis B or C
* CNS lymphoma
* previous malignancies, or cardiac, renal, hepatic, or respiratory failure
* Pregnant or lactating women and patients of child bearing potential unless using birth control measures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54
Dates: Start 2000-03; Study Completion 2006-08

PRIMARY OUTCOMES:
Toxicity during the treatment period
Efficacy evaluated in terms of complete and partial response 1 month after the end of therapy

SECONDARY OUTCOMES:
Efficacy evaluated in terms of molecular response ( bone marrow Bcl2 negativity after treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Sacchi Stefano, MD, Principal Investigator — GISL
Locations (9):
- Italy (9):
  - Ospedale di Arezzo, Arezzo
  - Ospedale Maggiore di Milano, Milan
  - Ospedale Monteluce, Perugia
  - Ospedale di Pescara, Pescara
  - Ospedale di Piacenza, Piacenza
  - Ospedale di Pisa, Pisa
  - Ospedale di Reggio Calabria, Reggio Calabria
  - Ospedale S. Maria Nuova, Reggio Emilia
  - Ospedale Molinette, Torino

REFERENCES:
- [Background] Alas S, Bonavida B. Rituximab inactivates signal transducer and activation of transcription 3 (STAT3) activity in B-non-Hodgkin's lymphoma through inhibition of the interleukin 10 autocrine/paracrine loop and results in down-regulation of Bcl-2 and sensitization to cytotoxic drugs. Cancer Res. 2001 Jul 1;61(13):5137-44. PMID 11431352
- [Background] Alas S, Emmanouilides C, Bonavida B. Inhibition of interleukin 10 by rituximab results in down-regulation of bcl-2 and sensitization of B-cell non-Hodgkin's lymphoma to apoptosis. Clin Cancer Res. 2001 Mar;7(3):709-23. PMID 11297268
- [Background] Di Gaetano N, Xiao Y, Erba E, Bassan R, Rambaldi A, Golay J, Introna M. Synergism between fludarabine and rituximab revealed in a follicular lymphoma cell line resistant to the cytotoxic activity of either drug alone. Br J Haematol. 2001 Sep;114(4):800-9. doi: 10.1046/j.1365-2141.2001.03014.x. PMID 11564066
- [Background] Bellosillo B, Villamor N, Colomer D, Pons G, Montserrat E, Gil J. In vitro evaluation of fludarabine in combination with cyclophosphamide and/or mitoxantrone in B-cell chronic lymphocytic leukemia. Blood. 1999 Oct 15;94(8):2836-43. PMID 10515887
- [Background] Sacchi S., Tucci A, Merli F, Orsucci L, Cervetti G, Occhini U, Liberati M, Tarantini G, Callea V, Brugiatelli M, Lauta VM, Baldini L, Luminari S, Federico M. Dipartimento di Oncologia ed Ematologia,. Phase II Study with Fludarabine and Cyclophosphamide Plus Rituximab (FC+R) in Relapsed Follicular Lymphoma Patients. ASH 2002. Blood 99, 2002 Ab n° 530
- See also: Related Info — http://www.gisl.org